CLINICAL TRIAL: NCT02283294
Title: Apixaban for Early Prevention of Recurrent Embolic Stroke and Hemorrhagic Transformation
Acronym: AREST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO00019754
Record Dates: First submitted 2014-10-29; First posted 2014-11-05 (Estimated); Results first posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2018-12

CONDITIONS: Transient Ischemic Attack; Stroke; Atrial Fibrillation
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke; Atrial Fibrillation | interventions — apixaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apixaban (Experimental): Apixaban twice a day for 180 days with drug initiation day 0-3 (TIA), day 3-5(small stroke) or day 7- 9 (medium stroke) respectively
  Interventions: Drug: Apixaban
- Warfarin (Active Comparator): standard of care warfarin starting at day 7±5 (TIA) or day 14 ±5 (small to medium ischemic stroke).
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Apixaban
  Arms: Apixaban
Drug: Warfarin
  Arms: Warfarin

SUMMARY:
The purpose of this study is to evaluate if Apixaban will decrease the complication of having another stroke for people who have atrial fibrillation if initiated earlier than standard of care.

DETAILED DESCRIPTION:
This is an Open label, randomized, active control, parallel-group pilot trial to examine the effect of initiation of APIXABAN at days 0-3 (TIA), days 3-5 (small stroke) and days 7-9 (medium stroke) to decrease fatal and/or recurrent stroke/TIA in 120 subjects who have suffered a recent( 0 to 48 hours from symptoms) TIA, or small to medium ischemic stroke compared to standard of care warfarin treatment regimen. Subjects will be randomly assigned in a 1:1 ratio to one of two treatment arms (apixaban or warfarin). Subjects will be followed for a total of 180 days during from screening through monthly follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent
2. Males and Females over 18 years of age.
3. History of Nonvalvular Atrial Fibrillation (NVAF) by documentation in the medical history or newly diagnosed nonvalvular Atrial Fibrillation at time of study randomization by ECG, device or telemetry .
4. Diagnosis of TIA or small or medium ischemic stroke 0 to 48 hours from signs or symptoms.
5. Women of child-bearing potential must use a reliable method of contraception and must provide a negative pregnancy test at entry into the study and within 24 hours of study treatment initiation.
6. WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug Apixaban plus 5 half-lives (approximately 3 days) plus 30 days (duration of ovulatory cycle) for a total of 33 days post-treatment completion.
7. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with Apixaban plus 5 half-lives (approximately 3 days) plus 90 days (duration of sperm turnover) for a total of 93 days post-treatment completion.
8. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However they must still undergo pregnancy testing as described in this section.

Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly.

At a minimum, subjects must agree to the use of one method of highly effective contraception as listed below:

HIGHLY EFFECTIVE METHODS OF CONTRACEPTION

* Male condoms with spermicide
* Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants and intrauterine devices (IUDs) such as Mirena by WOCBP subject or male subject's WOCBP partner. Female partners of male subjects participating in the study may use hormone based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug
* IUDs, such as ParaGard™
* Tubal ligation
* Vasectomy.
* Complete Abstinence

Exclusion Criteria:

1. Hemorrhagic stroke
2. Large ischemic stroke
3. History of major bleeding within the last 6 months from time of subject enrollment (e.g. GI bleed).
4. History of intracranial bleed

   a. Traumatic intracranial bleed within one year of randomization. (Traumatic ICH greater than one year of randomization is not an exclusion).
5. Current or history of bleeding disorders (e.g. blood dycrasias)
6. Blood Pressure of 180/100 mmHg on hypertensive therapy day of randomization per PI discretion 20.
7. Current illicit drug use and/or chronic alcohol use per PI discretion.
8. Severe liver disease (AST/ALT 2x upper limit).
9. Patients with kidney disease meeting criteria to take 2.5 mg twice daily who are taking strong dual inhibitors of CYP3A4 and P-glycoprotein (e.g. ketoconazole, itraconazole, ritonavir, clarithromycin) .
10. Any other suspected etiology for stroke (e.g. ipsilateral carotid disease).
11. Greater than 3 Cerebral Micro-bleeds (CMB) on gradient recovery echo (GRE) or evidence of intracranial hemorrhage on CT at time of randomization. (SWI sequencing may be used if GRE sequencing is not obtainable)
12. Therapeutically anti-coagulated at time of admission (INR at admission greater than 2.0 on warfarin or took two consecutive doses of NOAC).
13. Absolute indication for use of warfarin only.( e.g. Mechanical Valve)
14. Absolute indication for anticoagulation prior to randomization window. (e.g. DVT)
15. Hemoglobin less than 9 gm/dl and/or platelet count less than 100 K/uL.
16. Requires dual antiplatelet therapy.
17. Daily use of NSAIDS
18. Pregnancy or lactation.
19. Any use of an investigational product within the past 30 days.
20. Prisoners or subjects who are involuntarily incarcerated.
21. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
22. Concurrent participation in another clinical study where use of an investigational product is used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fradley, M.D., Principal Investigator — University of South Florida, Department of Cardiovascular Sciences
Locations (5):
- United States (5):
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Bayfront Health St Petersburg, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - University of Louisville, Louisville, Kentucky

REFERENCES:
- [Derived] Alrohimi A, Rose DZ, Burgin WS, Renati S, Hilker NC, Deng W, Oliveira GH, Beckie TM, Labovitz AJ, Fradley MG, Tran N, Gioia LC, Kate M, Ng K, Dowlatshahi D, Field TS, Coutts SB, Siddiqui M, Hill MD, Miller J, Jickling G, Shuaib A, Buck B, Sharma M, Butcher KS. Risk of hemorrhagic transformation with early use of direct oral anticoagulants after acute ischemic stroke: A pooled analysis of prospective studies and randomized trials. Int J Stroke. 2023 Aug;18(7):864-872. doi: 10.1177/17474930231164891. Epub 2023 Mar 26. PMID 36907985
- [Derived] Labovitz AJ, Rose DZ, Fradley MG, Meriwether JN, Renati S, Martin R, Kasprowicz T, Murtagh R, Kip K, Beckie TM, Stoddard M, Bozeman AC, McTigue T, Kirby B, Tran N, Burgin WS; AREST Investigators. Early Apixaban Use Following Stroke in Patients With Atrial Fibrillation: Results of the AREST Trial. Stroke. 2021 Apr;52(4):1164-1171. doi: 10.1161/STROKEAHA.120.030042. Epub 2021 Feb 25. PMID 33626904
- [Derived] Rose DZ, Meriwether JN, Fradley MG, Renati S, Martin RC, Kasprowicz T, Patel A, Mokin M, Murtagh R, Kip K, Bozeman AC, McTigue T, Hilker N, Kirby B, Wick N, Tran N, Burgin WS, Labovitz AJ. Protocol for AREST: Apixaban for Early Prevention of Recurrent Embolic Stroke and Hemorrhagic Transformation-A Randomized Controlled Trial of Early Anticoagulation After Acute Ischemic Stroke in Atrial Fibrillation. Front Neurol. 2019 Sep 20;10:975. doi: 10.3389/fneur.2019.00975. eCollection 2019. PMID 31620067

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ninety one patients were enrolled/consented into the study. Three patients of the 91 consented did not meet one or more of the inclusion/exclusion criteria and were excluded prior to randomization assignment.
Groups:
- Apixaban: Apixaban twice a day for 180 days with drug initiation day 0-3 (TIA), day 3-5(small stroke) or day 7- 9 (medium stroke) respectively
  Apixaban
- Warfarin: standard of care warfarin starting at day 7±5 (TIA) or day 14 ±5 (small to medium ischemic stroke).
  Warfarin
Period: Overall Study
Arm/Group | Apixaban | Warfarin
Started (Started indicates randomized to medication assignment. This does not necessarily indicate patient started the medication they were randomized to.) | 41 | 47
Received Allocated Treatment Intervention | 38 | 31
Completed | 38 | 39
Not Completed | 3 | 8
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 6
Not completed — Protocol Violation | 1 | 0
Not completed — Thrombus on transesophageal echocardiogram | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Warfarin | Total
Number analyzed (Participants) | 41 | 47 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 25
  >=65 years | 28 | 35 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.6 (14.9) | 74.3 (10.5) | 73.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 15 | 24 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 7 | 5 | 12
  Hispanic | 3 | 6 | 9
  Non-Hispanic White | 31 | 35 | 66
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 41 | 47 | 88
Hypertension [Count of Participants; unit: Participants] | 38 | 46 | 84
Hyperlipidemia [Count of Participants; unit: Participants] | 24 | 34 | 58
Coronary artery disease (CAD) [Count of Participants; unit: Participants] — Inclusive of history of untreated myocardial infarction, prior stenting, and prior coronary artery bypass graft. Does not include non-obstructive coronary disease.
  Participants | 13 | 18 | 31
Diabetes Mellitus [Count of Participants; unit: Participants] | 10 | 22 | 32
Peripheral Artery Disease [Count of Participants; unit: Participants] | 4 | 9 | 13
Prior Stroke [Count of Participants; unit: Participants] | 9 | 10 | 19
Prosthetic Heart Valve / Valve Replacement [Count of Participants; unit: Participants] | 1 | 4 | 5
Thyroid Disease [Count of Participants; unit: Participants] | 9 | 13 | 22
Obstructive Sleep Apnea [Count of Participants; unit: Participants] | 5 | 7 | 12
Congestive Heart Failure Symptoms [Count of Participants; unit: Participants] | 3 | 9 | 12
Past Medical History Left Ventricular Ejection Fraction < 40% [Count of Participants; unit: Participants] | 6 | 13 | 19
Chronic Kidney Disease Stage 3 [Count of Participants; unit: Participants] — glomerular filtration rate 30-59 mL/min/1.73 m^2
  Participants | 7 | 15 | 22
Chronic Kidney Disease Stage 4 [Count of Participants; unit: Participants] — glomerular filtration rate 15-29 mL/min/1.73 m^2
  Participants | 1 | 2 | 3
Chronic Kidney Disease Stage 5 [Count of Participants; unit: Participants] — glomerular filtration rate <15 or on dialysis
  Participants | 0 | 0 | 0
Transient Ischemic Attack [Count of Participants; unit: Participants] | 4 | 3 | 7
Thromboembolism History [Count of Participants; unit: Participants] | 0 | 3 | 3
New Onset Atrial Fibrillation [Count of Participants; unit: Participants] | 14 | 14 | 28
Prior Use of Anticoagulation within last 3 months [Count of Participants; unit: Participants] | 3 | 11 | 14
Former Tobacco Use History [Count of Participants; unit: Participants] | 10 | 13 | 23
Former Alcohol Use History [Count of Participants; unit: Participants] | 1 | 2 | 3
Former Illegal Drug Use History [Count of Participants; unit: Participants] | 1 | 1 | 2
Height [Mean (Standard Deviation); unit: m] | 1.67 (0.11) | 1.712 (0.14) | 1.69 (0.13)
Weight [Mean (Standard Deviation); unit: kg] | 82.10 (24.09) | 88.08 (24.73) | 85.29 (24.48)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.15 (6.68) | 30.05 (7.60) | 29.63 (7.16)
Body Surface Area [Mean (Standard Deviation); unit: m^2] | 1.90 (0.28) | 1.99 (0.31) | 1.95 (0.30)
Heart Rate [Mean (Standard Deviation); unit: bpm] | 76.56 (14.46) | 76.62 (16.61) | 76.60 (15.56)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 130.85 (18.64) | 134.53 (20.13) | 132.82 (19.43)
Current Tobacco Use [Count of Participants; unit: Participants] — Daily Use
  Participants | 0 | 4 | 4
Occasional Tobacco Use [Count of Participants; unit: Participants] — Less than daily user
  Participants | 0 | 0 | 0
Current Alcohol Use [Count of Participants; unit: Participants] — >/= 1 drink per day (1 drink = 12 ounces of regular beer, 5 ounces of wine, or 1.5 ounces of distilled spirits)
  Participants | 6 | 6 | 12
Occasional Alcohol Use [Count of Participants; unit: Participants] — <1 drink per day (1 drink = 12 ounces of regular beer, 5 ounces of wine, or 1.5 ounces of distilled spirits)
  Participants | 9 | 8 | 17
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 74.07 (17.76) | 70.26 (19.50) | 72.03 (18.70)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Composite Endpoint of Fatal Stroke, Recurrent Ischemic Stroke, or TIA
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 41 | 47
Participants | 7 | 12

2. Secondary Outcome: Number of Participants With an Intracranial Hemorrhage Assessed by MRI/CT
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 41 | 47
Participants | 5 | 6

ADVERSE EVENTS:
Time Frame: 210 +/- 10 days
Description: Adverse event assessment was performed at each of the patient follow up visits at baseline, day 14, day 30, day 60, day 120, day 150, day 180, and day 210. At each follow up visit, patients were evaluated by study coordinator, cardiologist, and neurologist. A physical exam, patient interview, electrocardiogram, and review of patient records were performed. Labs were evaluated for clinical significance at day 30, day 90, and day 180 visits.
Arm/Group | Apixaban | Warfarin
All-Cause Mortality (participants affected / at risk) | 2/41 | 4/47
Serious Adverse Events (participants affected / at risk) | 11/41 | 14/47
Other Adverse Events (participants affected / at risk) | 36/41 | 41/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=41) | Warfarin (N=47)
Pancreatic Cancer (Endocrine disorders) | 1 (1) | 0 (0)
Third Degree AV Block (Cardiac disorders) | 0 (0) | 2 (2)
Fatal Stroke (General disorders) | 1 (1) | 3 (3)
Worsening Congestive Heart Failure (Cardiac disorders) | 2 (2) | 0 (0)
Left Hip Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Worsening Atrial Fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Symptomatic Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Symptomatic PH1 Hemorrhagic Transformation (General disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TIA (General disorders) | 1 (1) | 2 (2)
GI Bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancolitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Acute Encephalopathy (General disorders) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Second Digit Right Foot Amputation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Recurrent Stroke (General disorders) | 5 (5) | 7 (7)
Back Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Worsening Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bilateral Leg Weakness / Trouble with Ambulation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Altered Mental Status (General disorders) | 0 (0) | 1 (1)
Metabolic Encephalopathy (General disorders) | 1 (1) | 0 (0)
Shortness of Breath (General disorders) | 0 (0) | 1 (1)
Symptomatic Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ostectomy Left Foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=41) | Warfarin (N=47)
Fatigue (Cardiac disorders) | 5 (5) | 5 (5)
Dizziness (Cardiac disorders) | 2 (2) | 9 (10)
Shortness of Breath (Cardiac disorders) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (6)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Intermittent Headaches (General disorders) | 5 (5) | 5 (5)
Urinary Tract Infection (Renal and urinary disorders) | 6 (6) | 3 (3)
Asymptomatic Bleed (General disorders) | 5 (5) | 5 (5)
Fever (General disorders) | 1 (1) | 0 (0)
Difficulty Finding Words (General disorders) | 2 (2) | 0 (0)
Intermittent Cognitive Impairment (General disorders) | 3 (3) | 2 (2)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Bilateral Lower Extremity Edema (Cardiac disorders) | 10 (11) | 3 (4)
Intermittent Leg Cramping (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Body / Muscle Aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Back Pain with Ambulation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cough (General disorders) | 2 (2) | 2 (3)
Dry Mouth (General disorders) | 1 (1) | 0 (0)
Altered Sense of Taste (General disorders) | 1 (1) | 1 (1)
Left Calf Sore (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Cold Symptoms (General disorders) | 1 (1) | 2 (2)
Sore Throat (General disorders) | 0 (0) | 1 (1)
Worsening Hearing Loss (General disorders) | 1 (1) | 0 (0)
Gout Right Foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Ataxia (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Right or Left Sided Weakness (General disorders) | 2 (2) | 1 (1)
Shakiness (General disorders) | 0 (0) | 1 (1)
Intermittent Lightheadedness (General disorders) | 2 (2) | 1 (1)
Blood Clot in Descending Aorta (Cardiac disorders) | 0 (0) | 1 (1)
Bronchitis (General disorders) | 3 (3) | 1 (1)
Pleuritic Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Decreased Appetite (Gastrointestinal disorders) | 0 (0) | 1 (1)
Generalized Weakness (General disorders) | 1 (1) | 1 (1)
Chest Pain or Tightness (Cardiac disorders) | 6 (6) | 3 (4)
Staph Infection Right Foot (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hemoptysis (General disorders) | 0 (0) | 1 (1)
Left Foot Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Intermittent Cardiac Pauses (Cardiac disorders) | 1 (1) | 0 (0)
Fall without Injury (Musculoskeletal and connective tissue disorders) | 7 (9) | 3 (3)
Left Foot Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Unsteady Gait (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intermittent Left Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Erectile Dysfunction (Renal and urinary disorders) | 1 (1) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Supratherapeutic INR (Cardiac disorders) | 0 (0) | 9 (29)
Left Eye Subconjunctival Hemorrhage (Eye disorders) | 0 (0) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 1 (2) | 8 (12)
Left Ankle Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vaginal Bleeding (Renal and urinary disorders) | 2 (3) | 0 (0)
Right Ankle Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 2 (2)
Hyponatremia (General disorders) | 0 (0) | 1 (1)
Right Foot Droop (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sensory Peripheral Neuropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fall with Injury (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Abrasions (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (8)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Orthostatic Loss of Consciousness (Cardiac disorders) | 1 (1) | 0 (0)
Acute Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypokalemia (General disorders) | 1 (1) | 0 (0)
Hyperkalemia (General disorders) | 1 (1) | 0 (0)
Facial and Neck Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Left Lower Facial Numbness (General disorders) | 1 (1) | 0 (0)
Nonsustained Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Bilateral Lower Extremity Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abnormal Liver Tests (Hepatobiliary disorders) | 1 (1) | 0 (0)
Parathesia (General disorders) | 1 (1) | 0 (0)
Total Bilirubin Elevated (Hepatobiliary disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Small Benign Cysts, Right Hepatic Lobe (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Muscle Spasticity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Upper Extremity Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Left Lower Extremity Edema (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertigo (General disorders) | 1 (1) | 0 (0)
Right Chest Basal Cell Removal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Upper Left Back Basal Cell Removal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Gastrointestinal Upset (Gastrointestinal disorders) | 0 (0) | 1 (1)
Left Middle Finger Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinus Infection (General disorders) | 0 (0) | 1 (1)
Bibasilar Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pacemaker Implant for Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Diaphoretic (General disorders) | 1 (1) | 0 (0)
Responsive Only to Painful Stimuli (General disorders) | 1 (1) | 0 (0)
Right Temporal Laceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Slurred Speech (General disorders) | 1 (1) | 0 (0)
Scalp Hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blood in Sputum (General disorders) | 0 (0) | 1 (1)
Minor Head Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right Great Toenail Removal Status Post Toe Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Left Hamstring Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Coarse Breath Sounds (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Actinic Keratosis Left Forearm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Squamous Cell Carcinoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Peeling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (2) | 0 (0)
Acute Gastric Ulcer with Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Diploplia (Eye disorders) | 0 (0) | 1 (1)
Blood in Semen (Renal and urinary disorders) | 0 (0) | 1 (1)
Abdominal Distention (Gastrointestinal disorders) | 0 (0) | 1 (2)
Motor Vehicle Accident with Injury (General disorders) | 0 (0) | 1 (1)
Right Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
White Tongue (General disorders) | 0 (0) | 1 (1)
Skin Lesion to Nose (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Generalized Body Numbness (General disorders) | 0 (0) | 1 (1)
Thrombus in Appendage (Cardiac disorders) | 0 (0) | 1 (1)
Syncopal Episode (General disorders) | 1 (1) | 0 (0)
Viral Illness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ear and Nose Infection (Infections and infestations) | 0 (0) | 1 (1)
Bladder Infection (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (1)
Midpelvic Mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fluid Overload (Cardiac disorders) | 0 (0) | 1 (1)
Heart Failure with Preserved Ejection Fraction (Cardiac disorders) | 0 (0) | 1 (1)
Right Lower Extremity Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bilateral Lower Extremity Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT02283294/Prot_SAP_000.pdf